CLINICAL TRIAL: NCT07393399
Title: Omega-3 Supplementation in Women With Systemic Lupus Erythematosus: Protocol for a Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Omega-3 Supplementation in Systemic Lupus Erythematosus
Acronym: SLE-OMEGA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Bruno Gualano, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: SLE_Omega3_RCT
Record Dates: First submitted 2026-01-30; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Lupus Erythematosus, Systemic
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omega-3 Supplementation (Experimental)
  Interventions: Dietary Supplement: Omega-3 Fatty Acids (EPA plus DHA)
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Omega-3 Fatty Acids (EPA plus DHA) — Oral omega-3 fatty acid supplementation (EPA+DHA), 5,400 mg/day for 12 weeks.
  Arms: Omega-3 Supplementation
Dietary Supplement: Placebo — Inert soybean oil capsules identical in appearance to the active supplement.
  Arms: Placebo

SUMMARY:
This randomized, double-blind, placebo-controlled clinical trial aims to evaluate whether oral omega-3 fatty acid supplementation can modulate inflammation, oxidative stress, and telomere maintenance in women with systemic lupus erythematosus (SLE) in remission. Women aged 18-45 years with SLE (SLEDAI-2K ≤ 4) will be allocated to receive either omega-3 (5,400 mg/day of EPA+DHA) or placebo for 12 weeks. A parallel healthy control group will undergo the same intervention scheme. Clinical, biochemical, and molecular assessments including inflammatory cytokines, oxidative stress markers (TBARS, ORAC, T-AOC), and relative telomere length (T/S ratio) will be conducted at baseline and post-intervention. The trial is designed to determine whether omega-3 can attenuate chronic low-grade inflammation and oxidative imbalance, both key drivers of cellular dysfunction and premature immunosenescence in SLE. Omega-3 PUFAs exert anti-inflammatory effects through competition with arachidonic acid for COX/LOX enzymes and by activating GPR120, which inhibits the TAK1-NF-κB-JNK inflammatory cascade. Their antioxidant effects may further reduce reactive oxygen species and support genomic stability. By integrating clinical, biochemical, and molecular outcomes, this study provides a comprehensive evaluation of omega-3 effects on pathways implicated in accelerated cellular aging in autoimmune diseases. The findings are expected to clarify whether omega-3 supplementation represents a safe, low-cost strategy capable of improving inflammatory and oxidative profiles and contributing to telomere preservation in women with SLE, supporting future precision-nutrition approaches in this population.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 to 45 years
* Diagnosis of systemic lupus erythematosus (SLE) according to the EULAR/ACR classification criteria
* Remission or low disease activity, defined as SLEDAI-2K ≤ 4
* On stable doses of hydroxychloroquine and/or glucocorticoids (≤10 mg/day of prednisone or equivalent) for at least 8 weeks prior to enrollment
* Ability and willingness to provide written informed consent
* Willingness to maintain usual dietary patterns and physical activity levels throughout the study period

Exclusion Criteria:

* Current use of omega-3 fatty acid supplements or use within the previous 3 months
* Pregnancy or lactation
* Presence of severe infection, neoplastic disease, or diabetes mellitus
* Known allergy or intolerance to fish oil or soybean oil
* Any medical condition or circumstance that, in the investigator's opinion, could interfere with study participation or adherence to the protocol

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 80 (Estimated)
Dates: Start 2026-07 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Telomere length | Baseline and 12 weeks
  Change in leukocyte telomere length assessed by quantitative polymerase chain reaction (qPCR), expressed as the telomere-to-single copy gene (T/S) ratio.

SECONDARY OUTCOMES:
Inflammatory markers | Baseline and 12 weeks
  Change in serum inflammatory markers, including interleukin-6 (IL-6) and high-sensitivity C-reactive protein (hs-CRP), assessed using standard laboratory methods.
Oxidative stress markers | Baseline and 12 weeks
  Change in oxidative stress markers, including malondialdehyde (MDA) and total antioxidant capacity (TAC), measured by validated biochemical assays.
Lipid profile | Baseline and 12 weeks
  Change in serum lipid profile, including total cholesterol, LDL-cholesterol, HDL-cholesterol, and triglycerides.

IPD SHARING:
Plan to Share IPD: Undecided